CLINICAL TRIAL: NCT00625313
Title: A Prospective, Multi-center, Single-phase, Non-randomized, Open-label Study to Assess the Safety and Efficacy of the HMY Model YA-60BB Intraocular Lens (IOL) for the Correction of Aphakia Following Phacoemulsification Cataract Extraction
Brief Title: Clinical Study of a UV-Absorbing Acrylic Posterior Chamber Intraocular Lens
Acronym: HMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoya Surgical Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSO 2003-A101
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Aphakia
Keywords: Cataract; aphakia; intraocular lens; IOL; Optical correction of aphakia
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HMY Model YA-60BB IOL (Experimental): Patients receiving a Hoya HMY Acrylic Foldable Intraocular Lens.
  Interventions: Device: HMY Model YA-60BB IOL

INTERVENTIONS:
Device: HMY Model YA-60BB IOL — Following phacoemulsification cataract extraction, insertion of a Hoya HMY posterior chamber intraocular lens will be performed.
  Other Names: Hoya HMY Acrylic Foldable Intraocular Lens

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the HMY Model YA-60BB Intraocular Lens (IOL) when implanted in the posterior chamber of the human eye for the optical correction of aphakia following cataract extraction.

DETAILED DESCRIPTION:
A prospective, single-phase, non-randomized, open-label study to include patients with operable cataract of the human crystalline lens who have a potential post-operative best corrected visual acuity of 20/40 or better and no pre-existing progressive sight-threatening ocular disorders. Patients who are eligible per inclusion / exclusion criteria will undergo phacoemulsification cataract extraction and then implantation of the Hoya HMY Model YA-60BB posterior chamber intraocular lens. Each patient will be followed-up at specific time intervals to assess safety and effectiveness, for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with cataract who are eligible for phacoemulsification cataract extraction of the lens through an incision of approximately 4 mm, and primary implantation of a posterior chamber intraocular lens.
2. Patients must have no pre-existing ocular conditions that preclude the ability of the treated eye to achieve BCVA of 20/40 or better after IOL implantation.
3. Patients must be at least 21 years of age.
4. Patients must sign a written informed consent form.
5. Patients must be able and willing to return for scheduled follow-up examinations after surgery throughout the 36 month study.

Exclusion Criteria:

1. Patients with a history of/or clinical signs of any of the following sight-threatening conditions:

   1. Previous Retinal Detachment or retinal pathology in operative eye, only
   2. Macular Degeneration in either eye
   3. Macular Edema in either eye
   4. Persistent Iritis/Uveitis in operative eye, only
2. Uncontrolled Glaucoma or under current treatment for glaucoma in either eye
3. Significant Corneal Disease in operative eye, only
4. Proliferative Diabetic Retinopathy in either eye
5. Patients who have had previous ocular surgery, of any kind, within the last 6 months or patients who have had previous ocular surgery at any time and who do not have potential BCVA after cataract extraction/IOL implantation of 20/40 or better
6. Patients who have best corrected vision worse than 20/200 in the fellow eye.
7. Patients with serious (i.e., life threatening) non-ophthalmic disease which may preclude study completion.
8. Patients who have undergone previous cataract extraction and intraocular lens implantation.
9. Patients unwilling or unable to sign the IRB-approved informed consent document for the study or who cannot or will not complete the study's examination schedule.
10. Patients who are currently enrolled in another clinical trial, or who exited a clinical trial within the last 30 days.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2004-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 12 months postoperative

SECONDARY OUTCOMES:
Adverse events/complications | 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Ziemba, M. Sc, Study Chair — Hoya Surgical Optics / Fullerton Regulatory & Clinical
Locations (1):
- Contact Hoya Surgical Optics, Inc. for Trial Locations, Chino Hills, California, United States